CLINICAL TRIAL: NCT01125228
Title: A Phase III Study With Long-Term Follow-Up of Zidovudine Versus Zidovudine and Alpha-Interferon Versus Alpha-Interferon in Patients With Early HIV Infection
Brief Title: Effectiveness of Zidovudine vs. Zidovudine Plus Alpha Interferon vs. Interferon for Treatment of HIV
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 880172; 88-I-0172
Record Dates: First submitted 2010-05-15; First posted 2010-05-18 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-08-19

CONDITIONS: HIV
Keywords: HIV; Natural History
MeSH Terms: interventions — Interferon-alpha

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AZT Alone: Zidovudine 200mg by mouth every 4hr
  Interventions: Drug: Ziodovudine and Alpha Interferon
- AZT plus IFN: -Zidovudine 200mg by mouth every 4hr -Alpha Interferon 1 million units once a day, escalating
  Interventions: Drug: Ziodovudine and Alpha Interferon
- IFN Alone: -Alpha Interferon 1 million units once a day, escalating

INTERVENTIONS:
Drug: Ziodovudine and Alpha Interferon
  Groups: AZT Alone; AZT plus IFN

SUMMARY:
This study will compare the effectiveness of zidovudine (AZT) alone vs. zidovudine plus interferon (IFN) vs. interferon alone in reducing HIV viral load, lessening immune system deterioration, and increasing the time to development of the first opportunistic infection in HIV-infected patients.

HIV-infected persons 18 years of age and older with a T4 lymphocyte count of 500/mm3 or more and no current opportunistic infections may be eligible for this study. Candidates will be screened with a medical history, physical examination, blood tests, chest X-ray, electrocardiogram, urinalysis, and, for patients with Kaposi s sarcoma lesions, measurement, photographs, and biopsy of lesions.

Patients will be assigned to receive treatment with either zidovudine alone, zidovudine plus interferon or interferon alone. They will continue treatment until one of the following occurs:

* Unacceptable side effects, despite dose modifications
* Development of an opportunistic infection
* Decrease in CD4 count by 20 percent or to an absolute count of less than 200/mm3
* Rapid progression of Kaposi s sarcoma lesions, requiring alternative therapy
* A decision is made to terminate the study

Patients will be followed long term for viral load, immune function, development of opportunistic infections, disease progression, and survival.

DETAILED DESCRIPTION:
Initial Study: THREE ARM (INTERVENTIONAL) STUDY

This randomized, controlled phase III protocol, initiated in 1988, was the first study to examine intervention with antiretroviral therapy and alpha interferon in patients with HIV infection. It evaluated the relative efficacy of zidovudine (AZT) vs. AZT + alpha interferon (IFN) vs. IFN in increasing time to first opportunistic infection, reducing HIV viremia, and lessening immune system deterioration in HIV-infected persons.

For the AZT alone arm, AZT dosing consisted of the standard regimen of 200 mg q4h. Persons on the AZT + IFN combination arm received AZT 100 mg q4h with IFN beginning at 1 million units qd, escalating up to 2.5 million units at 2 weeks, then in increments of 2.5 million units every 2 weeks. Patients on the IFN-alone arm began therapy at 5 million units qd and escalated in 2.5 million unit increments every 2 weeks, unless escalations were precluded by toxicity. Patients who had evidence of HIV infection and a CD4 countgreater than or equal to 500 were randomized to one of the three treatment groups. Patients were treated with their assigned medication until intolerable toxicity, opportunistic infection, or progressive Kaposi's sarcoma developed, or CD4 count declined to less than 200/mm(3).

Our statistically significant findings during this pre-HAART era study showed that interferon-alpha decreased HIV RNA viral load levels, both alone and in combination with AZT.

Long-Term Follow-up: EXTENSION PHASE (NATURAL HISTORY STUDY)

Once the intervention phase was completed, this protocol entered a long-term follow-up phase and evolved into a longitudinal natural history study. As of 2013, this work earned the distinction of following a cohort for 25 years or more. It continues to serve as an important source of data regarding the long-term outcomes of patients receiving anti-HIV treatment, and to provide information on the long-term consequences of therapy. In addition, stored blood and cells enable the study of cutting edge research questions, such as those related to immune activation, with new state-of-the-art laboratory assays.

ELIGIBILITY:
* INCLUSION CRITERIA:

Over 18 years of age.

T4 lymphocyte count greater than or equal to 500/mm3.

Infection with HIV as documented by positive ELISA and Western blot and positive HIV culture or positive p24 antigen or positive polymerase chain reaction.

Absence of current opportunistic infection (defined for purposes of this study as: candidiasis, cryptosporidiosis, mycobacterial infection, persistent herpes simplex infection, isosporiasis, cytomegalovirus infection, toxoplasmosis, pneumocystosis, salmonellosis, and cryptococcosis). Routine clinical methods and observations were performed to exclude such patients.

Afebrile (Temperature less the 38 degrees Centigrade orally) without antipyretics for at least 72 hours prior to enrollment.

Performance status 0, 1, or 2.

Relatively stable clinical condition, with no deterioration of performance status in the month prior to enrollment.

Ability to give informed consent and willing to comply with all procedures and visits scheduled.

Suitability of I.V. access for the scheduled blood tests.

Normal renal function as defined by BUN less than or equal to 30 and creatinine less than or equal to 1.5.

Normal hepatic function with transaminases and alkaline phosphatase less than 5 times the upper limit of normal range.

Hemoglobin greater than or equal to 10 gm/dl, total granulocyte count greater than or equal to 1250/mm(3), platelet count greater than or equal to 125,000/mm(3).

No previous therapy for KS within the month prior to enrollment, and no prior exposure to investigational agents. Prior exposure to AZT did not disqualify a patient; however patients were stratified on this basis.

EXCLUSION CRITERIA:

Patients with malignancy other than Kaposi's sarcoma were specifically excluded from this study.

Pregnant women, nursing mothers, or women of childbearing potential who were not employing effective means of contraception or abstinence.

Patients actively using illicit drugs.

Patients receiving systemically and potentially myelosuppressive drugs (such as TMP/SMX, pyrimethamine-sulfa or DHPG), nephrotoxic agents (such as amphotericin B or aminoglycosides), or cytotoxic or experimental chemotherapy.

Patients with a history of significant depressive disorder.

Patients with a history of an AIDS-defining opportunistic infection.

Subsequent Exclusion Criteria (Post Enrollment)

After enrollment, a patient was excluded from further participation in the study for any of the following reasons:

Serious infection not cleared by antibiotic therapy. The occurrence of a life-threatening infection, whether or not considered to be opportunistic, will prompt a discontinuation of therapy during the infection and for 2 weeks following its successful resolution. Therapy was re-initiated unless (1) in the investigator's judgment re-treatment with either or both of the study medications would be contraindicated for other reasons or (2) therapy had been held for more than 6 weeks.

Decrease in percent CD4 to less than 20 percent or in absolute CD4 count to less than 200/mm(3) on 3 consecutive blood tests.

Systemic allergic reaction to either study medication, characterized by angioedema, bronchial constriction, or anaphylaxis.

It was the principal investigator's judgment that the patient was too ill to continue in the trial.

Toxicity necessitating withdrawal.

Patient non-compliance: A patient not taking medication as directed or not keeping appointments was not allowed to continue on this study.

Rapid or life-threatening progression of KS such that the principal investigator believed other therapies would be in the patient's best interest.

Voluntary withdrawal: A patient could remove himself from study at any time. The patient was allowed to withdraw without prejudice.

Termination of the study by the principal investigator, sponsor, or the FDA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals infected with HIV during the 1980s and living throughout the US
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 1988-10-19 (Actual)

PRIMARY OUTCOMES:
Long term follow up | ongoing
  long-term follow-up of the medical and treatment outcomes of patients who received anti-HIV treatment and alpha-IFN in the pre-HAART era
sample collection | ongoing
  Ongoing prospective research plasma and cell collection as new lab assays and study questions continue to emerge (especially regarding immune activation and the pathways that drive it).

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Wright, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data related to the intervention phase of the study was already shared in published form in 2011: Tavel et al. https://www.liebertpub.com/doi/10.1089/jir.2009.0090 ). For the long-term observational follow-up phase of the study, individual data continues to be located in CRIMSON, CRIS, and Clinic 8 s Stored sample repository in Frederick. Participants signed consents allowing stored blood for future research for the duration of the protocol.
Supporting Information: Study Protocol
Time Frame: From start of study to present.
Access Criteria: Requests will be evaluated by the PI. Data will be shared if related to protocol objectives and will occur through encrypted, secure platforms. For NIH or outside investigator requests not related to protocol objectives, IRB approval will be required.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1988-I-0172.html